CLINICAL TRIAL: NCT06340516
Title: Monitoring Heart Function Through Blood Test Analysis of NT-proBNP During Treatment With HER2-Targeted Antibodies in HER2-Positive Breast Cancer - A Swedish Multicenter Study
Brief Title: NT-proBNP to Assess Trastuzumab-induced Cardiotoxicity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HER2BNP
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Cardiotoxicity; Breast Cancer; Treatment Side Effects
MeSH Terms: conditions — Cardiotoxicity; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a national multicentre phase II trial investigating the sensitivity and specificity of NT-proBNP for the diagnose of cardiac toxicity during primary anti-HER2 blockade. NT-proBNP is compared with the todays´ standard (ECHO/MUGA).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NT-proBNP instead of ECHO/MUGA at 6 months and 12 months (Experimental): Replacement with measurement of plasma levels of NT-proBNP at 6 months and 12 months instead of ECHO/MUGA for monitoring of trastuzumab-induced cardiotoxicity
  Interventions: Diagnostic Test: Plasma NT-proBNP

INTERVENTIONS:
Diagnostic Test: Plasma NT-proBNP — Replacement of measurement of plasma NT-proBNP instead of ECHO/MUGA at 6 months and 12 months of trastuzumab treatment to assess cardiotoxicity

SUMMARY:
Trastuzumab-induced cardiotoxicity (TIC) will be monitored in patients with HER2+ breast cancer undergoing trastuzumab treatment before and after breast cancer surgery. At baseline before start of trastuzumab treatment, echocardiography (ECHO)/multigated Acquisition Scan (MUGA) and measurement of plasma NT-proBNP will be performed. NT-proBNP will be measured again at 6 months and at 12 months of trastuzumab treatment. If elevations in NT-proBNP at 6 months and 12 months occur patients will be referred for ECHO/MUGA. The aim is to assess the sensitivity and specificity to detect TIC with NT-proBNP and whether ECHO/MUGA can be safely replaced by assessment of plasma NT-proBNP levels.

DETAILED DESCRIPTION:
Sponsor: Swedish Association of Breast Oncologists (SABO), Clinical Trial Unit, Department of Oncology, Sahlgrenska University Hospital, Gothenburg, Sweden.

Design:This is an national multicentre single arm phase II trial for patients with primary HER2 positive breast cancer planned for neoadjuvant/adjuvant treatment with HER2 blocking agents.

Purpose: The purpose of this study is to assess the sensitivity and specificity of NT-proBNP for detection of cardiac failure in patients with primary breast cancer that receive neoadjuvant/adjuvant treatment with HER2 blocking compounds.

Background: Patients with HER2 positive breast cancer > 20 mm and/or with lymph node metastasis receive, according to the national guidelines 4 courses of double antibody blockade with trastuzumab and pertuzumab plus a taxane for 12 weeks followed by EC (epirubicin/cyclophosphamide) every 3rd week times 3 in the neoadjuvant setting followed by continued HER2 blockade with trastuzumab or TDM-1 for a total of 17 courses. Patients with tumours < 20 mm and node-negative disease start with surgery followed by adjuvant treatment with EC x 4 followed by trastuzumab and a taxane for 12 weeks, thereafter trastuzumab x 13 is given as a single agent. For patients with tumours < 10 mm and node negative it is considered sufficient to give only a taxane plus trastuzumab for 12 weeks followed by trastuzumab times 13. The latter less toxic regimen has also been used in elderly fragile patients.

The risk of cardiac dysfunction as determined by a reduction in the Left Ventricular Ejection Fraction (LVEF) below 50% has been estimated to approximately 3-4% in the large registration trials.

Cardiac function is followed by repeated echocardiography (ECHO)/ Multigated Acquisition Scan (MUGA) that are performed before start of HER2 blocking treatment, after 6 and 12 months (when the treatment is completed.

Because cardiac toxicity is very low, a labour-intensive method needs to be carried out unnecessarily on a large number of patients. We have shown in a single centre pilot study of 136 patients that NT-proBNP has a high sensitivity and specificity compared with ECHO to correctly diagnose patients with cardiac toxicity during adjuvant/neoadjuvant HER2 treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmed HER2 positive primary BC planned for adjuvant/neoadjuvant treatment with chemotherapy plus HER2 blocking agents.
2. Patients ≥18 years
3. ECOG/WHO 0-1
4. Adequate organ function for the planned treatment according to local guidelines.
5. No distant metastasis (CT/MRI only if clinically indicated).
6. Negative pregnancy test within 14 days prior to start of treatment.
7. If of childbearing potential, willing to use an effective form of contraception.
8. No other malignancy during the last 5 years except for radically treated basal or squamous cell carcinoma of the skin or CIS of the cervix.
9. Signed informed consent and willingness to follow the trial procedures.

Exclusion Criteria:

1. Patients with previous heart disease recommended special follow-up during treatment with high risk of termination of treatment.
2. Evidence of any other medical conditions (such as psychiatric illness, infectious diseases, neurological conditions, physical examination or laboratory findings) that may interfere with the planned treatment or affect patient compliance.
3. Pregnancy and breast feeding.
4. Concurrent malignancy requiring therapy (excluding non-invasive carcinoma or carcinoma in situ).

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2029-03-14 (Estimated); Study Completion 2029-03-14 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of NT-proBNP to detect trastuzumab-induced cardiotoxicity | From inclusion to 24 months after baseline investigation
  To determine the sensitivity and specificity of NT-proBNP for identification of patients that develop cardiac toxicity during treatment with HER2 blocking agents for primary breast cancer [time frame from inclusion to 24 months after base-line investigation]

SECONDARY OUTCOMES:
Prevalence of trastuzumab-induced cardiotoxicity | From inclusion to 24 months after baseline investigation
  To determine the proportion of patients that develop cardiac toxicity during treatment with HER2 blocking agents for primary breast cancer
Anthracycline-induced change in NT-proBNP | From inclusion to 10 weeks after baseline investigation
  To investigate the potential change of NT-proBNP during anthracycline-based chemotherapy in patients that receive EC followed by anti-HER2 blockade plus a taxane and whether it is correlated with the development of cardiac toxicity throughout anti-HER2 blockade.
  [time frame from inclusion to 10 weeks after base-line investigation]

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Giglio, Assoc Prof, Principal Investigator — Sahlgrenska University Hospital/University of Gothenburg; Barbro Linderholm, Assoc Prof, Principal Investigator — Sahlgrenska University Hospital/University of Gothenburg
Locations (1):
- Jubileumskliniken, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No